CLINICAL TRIAL: NCT07302880
Title: The Acute Interference of Biotin in Blood Analysis
Acronym: ABBA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Nicolai Jacob Wewer Albrechtsen, Professor, MD, PhD, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ABBA
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Blood Sample; Interference With Routine Analyical Tests; Biotin Ingestion

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, cross-over study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Cohort A): 10 mg of biotin versus placebo (Experimental): Arm 1: 10 mg biotin → placebo (n = 6)
  Interventions: Other: Overall: To evaluate the acute effect of biotin intake on streptavidin-based laboratory assays during the hours immediately following consumption; Other: Arm 1 - 10 mg → Placebo
- Arm 2 (Cohort A): 10 mg of biotin versus placebo (Experimental): Arm 2: placebo → 10 mg biotin (n = 6)
  Interventions: Other: Overall: To evaluate the acute effect of biotin intake on streptavidin-based laboratory assays during the hours immediately following consumption; Other: Arm 2 - Placebo → 10 mg
- Arm 3 (Cohort B): 100 mg of biotin versus placebo (Experimental): Arm 3: 100 mg biotin → placebo (n = 6)
  Interventions: Other: Overall: To evaluate the acute effect of biotin intake on streptavidin-based laboratory assays during the hours immediately following consumption; Other: Arm 3 - 100 mg → Placebo
- Arm 4 (Cohort B): 100 mg of biotin versus placebo (Experimental): Arm 4: placebo → 100 mg biotin (n = 6)
  Interventions: Other: Overall: To evaluate the acute effect of biotin intake on streptavidin-based laboratory assays during the hours immediately following consumption; Other: Arm 4 - Placebo → 100 mg

INTERVENTIONS:
Other: Overall: To evaluate the acute effect of biotin intake on streptavidin-based laboratory assays during the hours immediately following consumption — The study will include two experimental days, each lasting 5 hours, as well as two short visits for a blood sample 24 hours after an experimental day.
  The setup is as follows:
  One study day with a single oral dose of biotin (randomized to either 10 mg or 100 mg), followed by a blood sample 24 hours after the study day with biotin.
  One study day with a single oral dose of placebo, followed by a blood sample 24 hours after the study day with placebo.
  The order of the two trials and the dose of biotin (either 10 mg or 100 mg) will also be randomized at inclusion.
  During the study day, subjects will rest in a supine position and an intravenous catheter is inserted into the left or right antecubital vein for collecting blood samples. Following a blood sample, subjects will receive an oral dose either 10 mg or 100 mg biotin or placebo. In total, blood will be sampled 8 times over a period of 5 hours. After 24 hours, the subject will visit again for a single blood sample.
Other: Arm 1 - 10 mg → Placebo — Participants receive a 10 mg oral dose of biotin on the first study day and placebo on the second study day. Blood samples are collected over 5 hours on each visit, with an additional fasting sample 24 hours later.
  Arms: Arm 1 (Cohort A): 10 mg of biotin versus placebo
Other: Arm 2 - Placebo → 10 mg — Participants receive placebo on the first study day and a 10 mg oral dose of biotin on the second study day. Blood samples are collected over 5 hours on each visit, with an additional fasting sample 24 hours later.
  Arms: Arm 2 (Cohort A): 10 mg of biotin versus placebo
Other: Arm 3 - 100 mg → Placebo — Participants receive a 100 mg oral dose of biotin on the first study day and placebo on the second study day. Blood samples are collected over 5 hours on each visit, with an additional fasting sample 24 hours later.
  Arms: Arm 3 (Cohort B): 100 mg of biotin versus placebo
Other: Arm 4 - Placebo → 100 mg — Intervention: Participants receive placebo on the first study day and a 100 mg oral dose of biotin on the second study day. Blood samples are collected over 5 hours on each visit, with an additional fasting sample 24 hours later.
  Arms: Arm 4 (Cohort B): 100 mg of biotin versus placebo

SUMMARY:
Biotin, also known as vitamin B7, is a water-soluble vitamin. It is essential for several metabolic processes in the body, including glucose, lipid, and protein metabolism, as it acts as a coenzyme in several carboxylation reactions. Biotin, available as an over the counter supplement, is widely used to improve nail and hair growth. The use of biotin supplements can interfere with various laboratory tests, due to the use of the streptavidin-biotin interaction in several immunoassays. We therefore wish to investigate acute impact of biotin supplementation on various laboratory assays, with focus on the immediate post-ingestion effects and the time frame in which biotin interference is most pronounced.

DETAILED DESCRIPTION:
Biotin, also known as vitamin B7, is a water-soluble vitamin. It is essential for several metabolic processes in the body, including glucose, lipid, and protein metabolism, as it acts as a coenzyme in several carboxylation reactions. Biotin, available as an over the counter supplement, is widely used to improve nail and hair growth. The use of biotin supplements can interfere with various laboratory tests, due to the use of the streptavidin-biotin interaction in several immunoassays. Therefore, if patients consume biotin supplements before blood tests, biotin may interfere with assays that rely on biotin-based analysis, especially in the first hours after biotin intake.

We therefore wish to investigate acute impact of biotin supplementation on various laboratory assays, with focus on the immediate post-ingestion effects and the time frame in which biotin interference is most pronounced.

This study will provide data crucial for developing guidelines to manage and interpret test results for patients who have recently taken biotin supplements.

The primary aim of this study is to evaluate the acute effect of biotin intake on streptavidin-based laboratory assays during the hours immediately following consumption.

The investigators hypothesize that biotin intake significantly affects the results of streptavidin-based laboratory assays for up to 5 hours after consumption, leading to inaccurate test results, and that the biotin interference subsides after 24 hours.

ELIGIBILITY:
Inclusion criteria:

* Male or female between 20-70 years of age at time of screening
* Body mass index of 18.6-25 kg/m2

Exclusion criteria:

* Severe liver disease (estimated by FIB4 score > 3.25)
* Type 2 diabetes according to ADA criteria (estimated by HbA1c levels of ≥ 48 mmol/mol)
* Significant history of alcoholism or drug/chemical abuse as per investigators judgement
* Kidney disease defined as serum creatinine levels ≥ 126 μmol/L for male and ≥ 111 μmol/L for female or eGFR < 60 ml/min/1.73 m2
* Cardiac problems (defined as troponin T levels > 10 ng/L for woman and >19 ng/L for men) or including any of the following, based on medical history:

  * Classified as being in New York Heart Association (NYHA) class III or IV
  * Angina pectoris (chest pain) within the last 6 months
  * Acute myocardial infarction (heart attack) within last 2 years
* Cancer within the past 1 year
* Anemia (hemoglobin <8.3 mmol/L for men and <7.3 mmol/L for women)
* Pregnancy (requires negative pregnancy test) or breast feeding
* Smoking
* Any medicine, acute illness (within the last two weeks) or other circumstances that in the opinion of the investigator might endanger the participants' safety or compliance with the protocol

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
The effect of 100 mg of biotin versus placebo on plasma levels of thyroid peroxidase antibody (TPOAb) | Blood sample on study day at timepoint = 120 minutes.
  The effect of 100 mg of biotin versus placebo on plasma levels of thyroid peroxidase antibody (TPOAb) (defined as the difference in peak concentration level of TPOAb at t=120 minutes, calculated as the fold change between study day with biotin (100 mg biotin) and study day with placebo).

SECONDARY OUTCOMES:
The effect of 100 mg of biotin versus placebo on plasma levels of thyroid peroxidase antibody (TPOAb) | Blood sample on study day at timepoint = 30, 60, 90, 180, 240, 300 minutes
  The effect of 100 mg of biotin versus placebo on plasma levels of thyroid peroxidase antibody (TPOAb) (defined as the difference in peak concentration level of TPOAb at t=30, 60, 90, 180, 240 and 300 minutes, calculated as the fold change between study day with biotin (100 mg biotin) and study day with placebo).
The effect of 10 mg of biotin versus placebo on plasma levels of thyroid peroxidase antibody (TPOAb) | Blood sample on study day at timepoint = 30, 60, 90, 120, 180, 240, 300 minutes
  The effect of 10 mg of biotin versus placebo on plasma levels of thyroid peroxidase antibody (TPOAb) (defined as the difference in peak concentration level of TPOAb at t= 30, 60, 90, 120, 180, 240 and 300, calculated as the fold change between study day with biotin (10mg biotin) and study day with placebo.)
The effect of 10 mg of biotin versus 100 mg biotin on plasma levels of thyroid peroxidase antibody (TPOAb) | Blood sample on study day at timepoint = 30, 60, 90, 120, 180, 240, 300 minutes
  The effect of 10 mg of biotin versus 100 mg biotin on plasma levels of thyroid peroxidase antibody (TPOAb) (defined as the difference in peak concentration level of TPOAb at t=30, 60, 90, 120, 180, 240 and 300 minutes, calculated as the fold change between study day with biotin (100 mg biotin) and study day with biotin (10 mg biotin).
The effect of 100 mg of biotin versus placebo on plasma levels of secondary outcomes | Blood sample on study day at timepoint = 30, 60, 90, 120, 180, 240, 300 minutes
  The effect of 100 mg of biotin versus placebo on plasma levels of secondary outcomes, including among others insulin, TSH, TnT, C-peptide, ProBNP (defined as the difference in peak concentration levels at t=30, 60, 90, 120, 180, 240 and 300 minutes, calculated as the fold change between study day with biotin (100 mg biotin) and study day with placebo).
The effect of 10 mg of biotin versus placebo on plasma levels of secondary outcomes | Blood sample on study day at timepoint = 30, 60, 90, 120, 180, 240, 300 minutes
  The effect of 10 mg of biotin versus placebo on plasma levels of secondary outcomes, including among others insulin, TSH, TnT, C-peptide, ProBNP (defined as the difference in peak concentration levels at t=30, 60, 90, 120, 180, 240 and 300 minutes, calculated as the fold change between study day with biotin (10 mg biotin) and study day with placebo).
The effect of 10 mg of biotin versus 100 mg on plasma levels of secondary outcomes | Blood sample on study day at timepoint = 30, 60, 90, 120, 180, 240, 300 minutes
  The effect of 10 mg of biotin versus 100 mg on plasma levels of secondary outcomes, including among others insulin, TSH, TnT, C-peptide, ProBNP (defined as the difference in peak concentration levels at t=30, 60, 90, 120, 180, 240 and 300 minutes, calculated as the fold change between study day with biotin (100 mg biotin) and study day with biotin (10 mg).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Biochemistry, Bispebjerg University Hospital, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
We have not decided to share IPD as this also would require approval from the ethical and data approval committee.